CLINICAL TRIAL: NCT04980391
Title: A Phase III, Double-blind, Randomized, Placebo-controlled Study to Evaluate the Safety, Reactogenicity and Immune Response of a Single Intramuscular Dose of Unadjuvanted RSV Maternal Vaccine, in High Risk Pregnant Women Aged 15 to 49 Years and Infants Born to the Vaccinated Mothers
Brief Title: A Study on the Safety and Immune Response to an Unadjuvanted RSV Maternal Vaccine, in High Risk Pregnant Women Aged 15 to 49 Years and Infants Born to the Vaccinated Mothers
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Following a recommendation from the Independent Data Monitoring Committee of NCT04605159 (RSV MAT 009), GSK made the decision to stop enrolment and vaccination in the study.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 214725; 2021-000994-96 (EudraCT Number)
Record Dates: First submitted 2021-07-20; First posted 2021-07-28 (Actual); Results first posted 2024-02-06 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-03

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: Respiratory Syncytial Virus Maternal vaccine; Safety; Reactogenicity; Immune response; High risk pregnant women; Teenage girls
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Masking Description: The study was unblinded to ensure the participant's safety.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- RSV_MAT Group (Experimental): Maternal participants randomized to the RSV_MAT Group received a single dose of the RSV MAT vaccine administered, between 24 and 36 weeks of gestation, at Day 1 in this study.
  Interventions: Biological: RSV MAT
- Control Group (Placebo Comparator): Maternal participants randomized to the Control Group received a single dose of Placebo administered, between 24 and 36 weeks of gestation, at Day 1 in this study.
  Interventions: Drug: Placebo
- RSV_MAT Group-Infant (No Intervention): This group consisted of infants born to mothers (from RSV_MAT Group-Mother) who received a single dose of RSV MAT vaccine during pregnancy.
- Control Group-Infant (No Intervention): This group consisted of infants born to mothers (from Control Group-Mother) who received a single dose of placebo during pregnancy.

INTERVENTIONS:
Biological: RSV MAT — Single dose of the RSV MAT vaccine reconstituted with NaCl solution, administered intramuscularly in the non-dominant arm, at Day 1.
  Arms: RSV_MAT Group
Drug: Placebo — Single dose of placebo, administered intramuscularly in the non-dominant arm, at Day 1.
  Arms: Control Group

SUMMARY:
The purpose of this study was to evaluate the safety, reactogenicity and immune response of a single intramuscular dose of the respiratory syncytial virus (RSV) maternal vaccine compared to placebo, when administered in the second or third trimester of pregnancy in women, 15 to 49 years of age (YOA), with high risk pregnancies and in the infants born to the vaccinated mothers.

Following a recommendation from the Independent Data Monitoring Committee of NCT04605159 (RSV MAT 009), GSK made the decision to stop enrolment and vaccination in the study. Ongoing study participants at that time continued to be monitored as part of the study.

ELIGIBILITY:
Inclusion Criteria:

Maternal participants

* Participants who can and will comply with the requirements of the protocol.
* Participants and LARs who give written or witnessed/thumb printed informed consent after the study has been explained according to local regulatory requirements, and before any study specific procedures are performed. The informed consent given at screening should either:

  * include consent for both the maternal participant's participation* and participation of the infant after the infant's birth, or
  * include consent for the maternal participant's participation* and expressed willingness to consider permitting the infant to take part after the infant's birth (if local regulations/guidelines require parent(s) to provide an additional informed consent after the infant's birth).
  * both mother and father should consent if local regulations / guidelines require it.
* Pre-pregnancy Body Mass Index (based on participant's report) 18.5 to 39.9 kg/m^2, inclusive.
* Healthy adolescent pregnant women, 15 to 17 YOA, inclusive, at the time of study intervention administration.

OR

* Pregnant women, 18 to 49 YOA, inclusive, at the time of study intervention administration with:

  * HIV infection AND/OR
  * Obstetric complications or risk factors during the current pregnancy, where the expectant management of the pregnancy is possible and without evidence of non-reassuring fetal status (only cases for which fetal heart rate can be ascertained) as follows:
  * Gestational diabetes, well-controlled on medications (with or without diet or exercise)
  * Gestational hypertension, well-controlled on diet or medications below 160/110 mmHg.
  * Pre-eclampsia without severe features (i.e. eclampsia, severe hypertension [>160/110 mmHg], organ dysfunction, unstable or complicated by [HELLP] syndrome).
  * Fetal Growth Restriction in singleton pregnancies, with normal umbilical artery Doppler and estimated fetal weight 3 to 10th percentile for gestational age.
  * History of threatened preterm labor in the current pregnancy, with no cervical dilation greater than 2 cm or effacement exceeding 50%, and/or no progressive change in cervical dilation or effacement detected by serial examinations, when maternal participant is asymptomatic
  * Uncomplicated twin gestation.
* Pregnant females at 24^0/7 to 36^0/7 weeks of gestation at the time of study intervention administration (Day 1), as established by:

  * Last menstrual period (LMP) date corroborated by first or second trimester ultrasound examination (U/S) (i.e. at or before 28 weeks of gestation).
  * First or second trimester U/S only, if LMP is unknown/uncertain.
  * Certain LMP, corroborated by an U/S performed after 28 weeks of gestation is also acceptable.

The level of diagnostic certainty of the gestational age should be established by using the Global Alignment of Immunization Safety Assessment in pregnancy (GAIA) gestation age assessment tool

* Participants who are willing to provide cord blood.
* Willing to have their offspring followed-up after delivery for a period of 12 months.
* Participants who do not plan to give their offspring for adoption or place the child in care.

Note that women whose pregnancies resulted from Assisted Reproductive Technologies may be enrolled if they meet all inclusion criteria and none of the exclusion criteria.

Infant participants

* Live-born from the study pregnancy.
* If required per local regulations / guidelines, re-signed (confirmed) written or witnessed/thumb printed informed consent for study participation of the infant obtained from the infant's mother and/or father and/or LAR, before performing any infant study specific procedure. To comply with RTI surveillance and other protocol required procedures that begin immediately after birth: if written consent cannot be provided by the parent(s)/LAR(s) readily post-birth, verbal consent - if permitted per local regulation -- may be sought from the parent(s) / LAR(s) instead. Verbal consent should be documented in the source data by the investigator or delegate. The parent(s) / LAR(s) will provide additional, written informed consent by (or before) Visit 2-NB.

Exclusion Criteria:

Maternal participants Medical conditions

* History of any reaction or hypersensitivity likely to be exacerbated by any component of the study intervention.
* Hypersensitivity to latex.
* Any pre-existing medical conditions or obstetric complications in the current pregnancy that, are poorly controlled and/or with clinical evidence of a non-reassuring fetal status and/or are likely to result in delivery within 7 days after study intervention administration and/or when the timing of planned delivery is within 7 days after study intervention administration and/or acute conditions requiring immediate medical attention for maternal stabilization and/or treatment.
* A multiple pregnancy with 3 or more fetuses.
* Complicated twin gestation.
* Placenta Accreta Spectrum, including placenta increta, percreta, and accreta.
* Fetal structural defects or genetic abnormalities that affect (or are likely to affect) fetal health or survival during the first year of life.
* Known or suspected impairment of the immune system or immunodeficiency syndrome other than HIV.
* Lymphoproliferative disorder or malignancy within 5 years before study dose administration.
* Any illness of the mother or conditions of the fetus that, may substantially interfere with the maternal participant's ability to comply with study procedures, or could increase the risks to the mother or the fetus, or could preclude the evaluation of the participant's data.
* Any other clinical condition that, might pose additional risk to the participant due to participation in the study, as determined by medical history, physical examination or laboratory screening tests.
* Women with any diagnosis, condition, treatment, or other factor that, has the potential to affect or confound assessments of immunogenicity or safety
* Any conditions which, in the investigator's opinion, would increase the risks of study participation to the unborn infant.

Prior/Concomitant therapy

* Prior receipt of an RSV maternal vaccine.
* Use of any investigational or non-registered product other than the study intervention(s) during the period beginning:

  * For a drug, vaccine or medical device: 29 days before the dose of study intervention(s) (Day -28 to Day 1), or their planned use during the study period.
  * For immunoglobulins: 90 days before the dose of study intervention(s), or their planned use during the study period.

The exception to this is investigational products administered in the setting of a pandemic. Administration in this case should respect the same period outlined above prior to study intervention administration, but may be allowed following delivery.

* Planned administration/administration of a vaccine not foreseen by the study protocol in the period starting 29 days before the study Day 1 and ending at delivery, with the exception of seasonal influenza vaccines, tetanus vaccines, dTpa/Tdap - alone vaccines, dTpa/Tdap vaccines that also contain other antigens and Hepatitis B vaccines, all of which may be administered according to standard of care ≥ 15 days before or after study intervention (Day 1).
* Receipt of blood or plasma products or immunoglobulin, from 90 days before study intervention administration, or planned receipt through delivery, with the exception of Rho(D) immunoglobulin, which can be given at any time. In that sense, COVID-19 vaccines may be allowed, when administered ≥ 15 days before or after study vaccination.
* Administration of immune-modifying therapy within 6 months before study intervention administration, or planned administration through delivery, except if it is part of management of HIV infection.

Prior/Concurrent clinical study experience

• Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational intervention.

Other exclusions

* Alcoholism or substance use disorder within the past 24 months based on the presence of 2 or more of the following abuse criteria: hazardous use, social/interpersonal problems related to use, neglect of major roles to use, withdrawal, tolerance, use of larger amounts or longer, repeated attempts to quit or control use, much time spent using, physical or psychological problems related to use, activities given up to use, craving.
* A local condition that precludes injection of the study vaccine/product or precludes assessment of local (administration site) reactogenicity.
* Consanguinity of maternal participant and her partner.
* Any study personnel or their immediate dependents, family, or household members.

Infant participants

* Concurrently participating in another clinical trial, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational vaccine/product.
* Any condition which, would increase the risks of study participation to the infant.
* Child in care.

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Only pregnant women, 15 to 49 YOA were included in the study.
Enrollment: 384 (Actual)
Dates: Start 2021-08-03 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (33):
- United States (16):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Dothan, Alabama
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Covington, Louisiana
  - GSK Investigational Site, Lafayette, Louisiana
  - GSK Investigational Site, Slidell, Louisiana
  - GSK Investigational Site, Missoula, Montana
  - GSK Investigational Site, Arlington, Texas
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Grapevine, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, League City, Texas
  - GSK Investigational Site, Plano, Texas
  - GSK Investigational Site, Weatherford, Texas
- Brazil (3):
  - GSK Investigational Site, Caxias do Sul
  - GSK Investigational Site, RibeirAo PretoSP
  - GSK Investigational Site, Santa Maria
- Canada (2):
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Montreal, Quebec
- GSK Investigational Site, Helsinki, Finland
- India (2):
  - GSK Investigational Site, Bhubaneswar
  - GSK Investigational Site, Mysuru
- Italy (3):
  - GSK Investigational Site, Messina
  - GSK Investigational Site, Perugia
  - GSK Investigational Site, Prato
- GSK Investigational Site, Panama City, Panama
- GSK Investigational Site, Soweto Gauteng, South Africa
- Spain (4):
  - GSK Investigational Site, Boadilla Del Monte Madrid
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, TorrejOn Ardoz Madrid

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 384 participants who completed the informed consent process, 169 maternal participants were vaccinated, and 198 infants, including twins, were born to those exposed mothers (RSV_MAT Group-Mother and Control Group-Mother). Therefore, 367 participants were considered exposed.
Groups:
- RSV_MAT Group-Mother: Maternal participants randomized to the RSV_MAT Group received a single dose of the RSV MAT vaccine administered, between 24 and 36 weeks of gestation, at Day 1 in this study.
- Control Group-Mother: Maternal participants randomized to the Control Group received a single dose of Placebo administered, between 24 and 36 weeks of gestation, at Day 1 in this study.
Period: Overall Study
Arm/Group | RSV_MAT Group-Mother | Control Group-Mother | RSV_MAT Group-Infant | Control Group-Infant
Started | 113 | 56 | 132 | 66
Completed | 107 | 52 | 124 | 61
Not Completed | 6 | 4 | 8 | 5
Not completed — Death | 0 | 0 | 1 | 1
Not completed — Lost to Follow-up | 3 | 3 | 2 | 3
Not completed — WITHDRAWAL BY SUBJECT, NOT DUE TO AN ADVERSE EVENT | 2 | 0 | 0 | 0
Not completed — MIGRATED / MOVED FROM THE STUDY AREA | 1 | 1 | 2 | 1
Not completed — WITHDRAWAL BY SUBJECT'S PARENT(S)/LAR(S) | 0 | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RSV_MAT Group-Mother | Control Group-Mother | RSV_MAT Group-Infant | Control Group-Infant | Total
Number analyzed (Participants) | 113 | 56 | 132 | 66 | 367
Age, Customized [Count of Participants; unit: Participants]
  0 to 1 years of age | 0 | 0 | 132 | 66 | 198
  15 < 18 years of age | 13 | 6 | 0 | 0 | 19
  18 to 49 years of age | 100 | 50 | 0 | 0 | 150
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113 | 56 | 63 | 29 | 261
  Male | 0 | 0 | 69 | 37 | 106
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 4 | 1 | 4 | 1 | 10
  Black or African American | 33 | 18 | 33 | 18 | 102
  White | 52 | 24 | 67 | 34 | 177
  Other, unspecified | 24 | 13 | 28 | 13 | 78

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Maternal Participants Reporting Any Solicited Administration Site Events
Description: Assessed solicited administration site events included erythema, pain and swelling. Any pain = occurrence of the symptom regardless of intensity grade. Any erythema and swelling = symptom reported with a surface diameter greater than or equal to 20 millimeters.
Time Frame: From Day 1 to Day 7 included
Population: Analysis was performed on the Solicited Safety Set, which included all maternal participants who received 1 dose of a study intervention and who had solicited safety data available during the specified period.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RSV_MAT Group-Mother | Control Group-Mother
Number analyzed (Participants) | 113 | 54
Percentage of participants
  Any Erythema | 0.9 [0.0 to 4.8] | 0 [0 to 6.6]
  Any Pain | 44.2 [34.9 to 53.9] | 14.8 [6.6 to 27.1]
  Any Swelling | 0 [0 to 3.2] | 1.9 [0.0 to 9.9]

2. Primary Outcome: Percentage of Maternal Participants Reporting Any Solicited Systemic Events
Description: Assessed solicited systemic events included abdominal pain, diarrhea, fatigue, headache, nausea, fever [temperature equal to or above (>=) 38 degrees Celsius (°C)/100.4 degrees Fahrenheit (°F), regardless of the location of measurement] and vomiting. Any = occurrence of the adverse event regardless of intensity grade or relation to study vaccination.
Time Frame: From Day 1 to Day 7 included
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RSV_MAT Group-Mother | Control Group-Mother
Number analyzed (Participants) | 113 | 54
Percentage of participants
  Any Abdominal pain | 20.4 [13.4 to 29.0] | 16.7 [7.9 to 29.3]
  Any Diarrhea | 20.4 [13.4 to 29.0] | 7.4 [2.1 to 17.9]
  Any Fatigue | 28.3 [20.2 to 37.6] | 27.8 [16.5 to 41.6]
  Any Headache | 39.8 [30.7 to 49.5] | 38.9 [25.9 to 53.1]
  Any Nausea | 24.8 [17.1 to 33.8] | 20.4 [10.6 to 33.5]
  Any Fever | 0 [0 to 3.2] | 0 [0 to 6.6]
  Any Vomiting | 8.0 [3.7 to 14.6] | 20.4 [10.6 to 33.5]

3. Primary Outcome: Percentage of Maternal Participants Reporting Any Unsolicited Adverse Events (AEs)
Description: An unsolicited AE was defined as any AE reported in addition to those solicited during the clinical study. Also, any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms was reported as an unsolicited AE. Any = occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: From Day 1 to Day 30 included
Population: Analysis was performed on the Exposed Set - Maternal, which included all maternal participants who received 1 dose of a study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RSV_MAT Group-Mother | Control Group-Mother
Number analyzed (Participants) | 113 | 56
Percentage of participants | 34.5 [25.8 to 44.0] | 37.5 [24.9 to 51.5]

4. Primary Outcome: Percentage of Maternal Participants Reporting Any Serious Adverse Events (SAEs) From Day 1 up to 42 Days Post-delivery
Description: An SAE was defined as any untoward medical occurrence that resulted in death, was life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity, was a congenital anomaly/birth defect in the offspring of a study participant or resulted in abnormal pregnancy outcomes or in other situations that were considered serious per medical or scientific judgment. Any = occurrence of any SAE regardless of intensity grade or relation to vaccination.
Time Frame: From Day 1 up to 42 days post-delivery, an average of 2 months
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RSV_MAT Group-Mother | Control Group-Mother
Number analyzed (Participants) | 113 | 56
Percentage of participants | 29.2 [21.0 to 38.5] | 19.6 [10.2 to 32.4]

5. Primary Outcome: Number of Maternal Participants Reporting (S)AEs Leading to Study Withdrawal From Day 1 up to 42 Days Post-delivery
Description: A participant was considered to have withdrawn from the study if no new study procedure had been performed or no new information had been collected for her since the date of withdrawal/last contact. (S)AEs leading to study withdrawal were (S)AEs identified by the investigator to cause participant withdrawal until the resolution of the event. These participant withdrawals were considered different from participant withdrawals for other reasons.
Time Frame: From Day 1 up to 42 days post-delivery, an average of 2 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | RSV_MAT Group-Mother | Control Group-Mother
Number analyzed (Participants) | 113 | 56
Participants | 0 | 0

6. Primary Outcome: Percentage of Maternal Participants Reporting Medically Attended Adverse Events (MAEs) From Day 1 up to 42 Days Post-delivery
Description: An MAE was defined as an unsolicited AE for which the participant received medical attention such as hospitalization, or an emergency room visit, or visit to/by a health care provider.
Time Frame: From Day 1 up to 42 days post-delivery, an average of 2 months
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RSV_MAT Group-Mother | Control Group-Mother
Number analyzed (Participants) | 113 | 56
Percentage of participants | 57.5 [47.9 to 66.8] | 58.9 [45.0 to 71.9]

7. Primary Outcome: Percentage of Live Births With no Congenital Anomalies, Live Births With Minor Congenital Anomaly(Ies) and Live Births With at Least 1 Major Congenital Anomaly
Description: The percentage of live births with no congenital anomalies, live births with minor congenital anomaly(ies) only and live births with at least 1 major congenital anomaly is reported.
Time Frame: From Day 1 up to 42 days post-delivery, an average of 2 months
Population: Analysis was performed on the Exposed Set - Infant, which included infants live-born to exposed maternal participants, whose parents/legally acceptable representatives (LARs) completed the informed consent process and signed the informed consent form.
Measure: Number (95% Confidence Interval); unit: Percentage of live births
Arm/Group | RSV_MAT Group-Infant | Control Group-Infant
Number analyzed (Participants) | 132 | 66
Percentage of live births
  LIVE BIRTH WITH NO CONGENITAL ANOMALIES | 86.4 [79.3 to 91.7] | 84.8 [73.9 to 92.5]
  LIVE BIRTH WITH ONLY MINOR CONGENITAL ANOMALY(IES) | 10.6 [5.9 to 17.2] | 13.6 [6.4 to 24.3]
  LIVE BIRTH WITH AT LEAST ONE MAJOR CONGENITAL ANOMALY | 3.0 [0.8 to 7.6] | 1.5 [0.0 to 8.2]

8. Primary Outcome: Percentage of Maternal Participants Reporting Pregnancy-related Adverse Events of Special Interest (AESIs) From Day 1 up to 42 Days Post-delivery
Description: Pregnancy-related AESIs included preterm labor, provider-initiated preterm birth, premature preterm rupture of membranes, pre-eclampsia, pre-eclampsia with severe features including eclampsia, gestational hypertension and fetal growth restriction.
Time Frame: From Day 1 up to 42 days post-delivery, an average of 2 months
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RSV_MAT Group-Mother | Control Group-Mother
Number analyzed (Participants) | 113 | 56
Percentage of participants
  Preterm labor | 8.0 [3.7 to 14.6] | 7.1 [2.0 to 17.3]
  Provider-initiated preterm birth | 3.5 [1.0 to 8.8] | 5.4 [1.1 to 14.9]
  Premature preterm rupture of membranes | 1.8 [0.2 to 6.2] | 5.4 [1.1 to 14.9]
  Pre-eclampsia | 4.4 [1.5 to 10.0] | 3.6 [0.4 to 12.3]
  Pre-eclampsia with severe features including eclampsia | 4.4 [1.5 to 10.0] | 0 [0 to 6.4]
  Gestational hypertension | 0.9 [0.0 to 4.8] | 3.6 [0.4 to 12.3]
  Fetal growth restriction | 1.8 [0.2 to 6.2] | 3.6 [0.4 to 12.3]

9. Primary Outcome: Percentage of Maternal Participants Reporting Worsening of Pre-existing Medical Conditions and/or Obstetric Complications From Day 1 up to 42 Days Post-delivery
Description: Worsening of pre-existing medical condition and/or obstetric complication was considered by the investigator, using clinical judgment and the following criteria:
  * Change in medication and/or medication dose.
  * Medically attended event in relation to pre-existing condition and/or obstetric complication that are outside the routine management of the condition/complication.
  * SAE and/or hospitalization in relation to pre-existing condition and/or obstetric complication.
Time Frame: From Day 1 up to 42 days post-delivery, an average of 2 months
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RSV_MAT Group-Mother | Control Group-Mother
Number analyzed (Participants) | 113 | 56
Percentage of participants
  Change In Medication And/Or Medication Dose | 1.8 [0.2 to 6.2] | 1.8 [0.0 to 9.6]
  Medically Attended Event In Relation To Pre-Existing Condition And/Or Obstetric Complication | 1.8 [0.2 to 6.2] | 7.1 [2.0 to 17.3]
  SAE And/Or Hospitalization In Relation To Pre-Existing Condition And/Or Obstetric Complication | 1.8 [0.2 to 6.2] | 3.6 [0.4 to 12.3]

10. Primary Outcome: Percentage of Infant Participants Reporting Neonatal/Infant AESIs From Birth up to 42 Days Post-birth
Description: Neonatal/infant AESIs included low birth weight (below [<] 2500 grams), very low birth weight (<1500 grams), extremely low birth weight (<1000 grams), preterm birth (<37 weeks of gestational age), small for gestational age (weight below 10th percentile for gestational age), congenital anomalies with internal structural defects and neonatal death in a preterm live birth (gestational age equal to or above [>=] 28 and <37 weeks).
Time Frame: From birth up to 42 days post-birth, an average of 2 months
Population: Analysis was performed on the Exposed Set - Infant, which included infants live-born to exposed maternal participants, whose parents/LARs completed the informed consent process and signed the informed consent form.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RSV_MAT Group-Infant | Control Group-Infant
Number analyzed (Participants) | 132 | 66
Percentage of participants
  Low Birth Weight (<2500 grams) | 16.7 [10.7 to 24.1] | 18.2 [9.8 to 29.6]
  Very Low Birth Weight (<1500 grams) | 2.3 [0.5 to 6.5] | 1.5 [0.0 to 8.2]
  Extremely Low Birth Weight (<1000 grams) | 0 [0 to 2.8] | 1.5 [0.0 to 8.2]
  Preterm Birth (<37 Weeks Of Gestational Age) | 18.2 [12.0 to 25.8] | 19.7 [10.9 to 31.3]
  Small For Gestational Age | 14.4 [8.9 to 21.6] | 27.3 [17.0 to 39.6]
  Congenital Anomalies With Internal Structural Defects | 3.0 [0.8 to 7.6] | 0 [0 to 5.4]
  Neonatal Death In A Preterm Live Birth (gestational age >=28 and <37 weeks) | 0.8 [0.0 to 4.1] | 1.5 [0.0 to 8.2]

11. Primary Outcome: Percentage of Infant Participants Reporting Any SAEs From Birth up to 42 Days Post-birth
Description: An SAE was defined as any untoward medical occurrence that resulted in death, was life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity, was a congenital anomaly/birth defect or resulted in other situations that were considered serious per medical or scientific judgment. Any = occurrence of any SAE regardless of intensity grade or relation to vaccination.
Time Frame: From birth up to 42 days post-birth, an average of 2 months
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RSV_MAT Group-Infant | Control Group-Infant
Number analyzed (Participants) | 132 | 66
Percentage of participants | 20.5 [13.9 to 28.3] | 27.3 [17.0 to 39.6]

12. Primary Outcome: Number of Infant Participants Reporting (S)AEs Leading to Study Withdrawal From Birth up to 42 Days Post-birth
Description: as for outcome 5
Time Frame: From birth up to 42 days post-birth, an average of 2 months
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | RSV_MAT Group-Infant | Control Group-Infant
Number analyzed (Participants) | 132 | 66
Participants | 0 | 0

13. Primary Outcome: Percentage of Infant Participants Reporting MAEs From Birth up to 42 Days Post-birth
Description: An MAE was defined as an unsolicited AE for which the participants received medical attention such as hospitalization, or an emergency room visit, or visit to/by a health care provider.
Time Frame: From birth up to 42 days post-birth, an average of 2 months
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RSV_MAT Group-Infant | Control Group-Infant
Number analyzed (Participants) | 132 | 66
Percentage of participants | 56.8 [47.9 to 65.4] | 54.5 [41.8 to 66.9]

14. Primary Outcome: Percentage of Infant Participants Reporting Any SAEs From Birth up to 180 Days Post-birth
Description: as for outcome 11
Time Frame: From birth up to 180 days post-birth
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RSV_MAT Group-Infant | Control Group-Infant
Number analyzed (Participants) | 132 | 66
Percentage of participants | 25.0 [17.9 to 33.3] | 30.3 [19.6 to 42.9]

15. Primary Outcome: Number of Infant Participants Reporting (S)AEs Leading to Study Withdrawal From Birth up to 180 Days Post-birth
Description: as for outcome 5
Time Frame: From birth up to 180 days post-birth
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | RSV_MAT Group-Infant | Control Group-Infant
Number analyzed (Participants) | 132 | 66
Participants | 0 | 0

16. Primary Outcome: Percentage of Infant Participants Reporting MAEs From Birth up to 180 Days Post-birth
Description: as for outcome 13
Time Frame: From birth up to 180 days post-birth
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RSV_MAT Group-Infant | Control Group-Infant
Number analyzed (Participants) | 132 | 66
Percentage of participants | 77.3 [69.2 to 84.1] | 69.7 [57.1 to 80.4]

17. Primary Outcome: Percentage of Infant Participants Reporting Any SAEs From Birth up to 365 Days Post-birth
Description: as for outcome 11
Time Frame: From birth up to 365 days post-birth
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RSV_MAT Group-Infant | Control Group-Infant
Number analyzed (Participants) | 132 | 66
Percentage of participants | 26.5 [19.2 to 34.9] | 31.8 [20.9 to 44.4]

18. Primary Outcome: Number of Infant Participants Reporting (S)AEs Leading to Study Withdrawal From Birth up to 365 Days Post-birth
Description: as for outcome 5
Time Frame: From birth up to 365 days post-birth
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | RSV_MAT Group-Infant | Control Group-Infant
Number analyzed (Participants) | 132 | 66
Participants | 0 | 0

19. Primary Outcome: Percentage of Infant Participants Reporting MAEs From Birth up to 365 Days Post-birth
Description: as for outcome 13
Time Frame: From birth up to 365 days post-birth
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RSV_MAT Group-Infant | Control Group-Infant
Number analyzed (Participants) | 132 | 66
Percentage of participants | 86.4 [79.3 to 91.7] | 75.8 [63.6 to 85.5]

20. Primary Outcome: RSV MAT Immunoglobulin G (IgG)-Specific Antibody Concentrations for Maternal Participants at Pre-dosing (Day 1)
Description: RSV MAT IgG-specific antibody concentrations were determined by enzyme-linked immunosorbent assay (ELISA) and expressed as geometric mean concentrations (GMCs) in ELISA units per milliliter (ELU/mL).
Time Frame: At pre-dosing (Day 1)
Population: Analysis was performed on the Per Protocol Set Immunogenicity - Maternal, which included all maternal participants who received 1 dose of a study intervention and had immunogenicity data available for the specified analysis at the specified time point (i.e. pre-dosing [Day 1]), minus those participants with protocol deviations that lead to exclusion.
Measure: Geometric Mean (95% Confidence Interval); unit: ELU/mL
Arm/Group | RSV_MAT Group-Mother | Control Group-Mother
Number analyzed (Participants) | 103 | 48
ELU/mL | 4981.6 [4405.14 to 5633.53] | 5981.7 [4908.71 to 7289.11]

21. Primary Outcome: RSV MAT IgG-specific Antibody Concentrations for Maternal Participants at Delivery
Description: RSV MAT IgG-specific antibody concentrations were determined by ELISA and expressed as GMCs in ELU/mL.
Time Frame: At delivery
Population: Analysis was performed on the Per Protocol Set Immunogenicity - Maternal, which included all maternal participants who received 1 dose of a study intervention and had immunogenicity data available for the specified analysis at the specified time point (i.e. delivery), minus those participants with protocol deviations that lead to exclusion.
Measure: Geometric Mean (95% Confidence Interval); unit: ELU/mL
Arm/Group | RSV_MAT Group-Mother | Control Group-Mother
Number analyzed (Participants) | 99 | 44
ELU/mL | 70337.1 [60711.34 to 81489.07] | 4421 [3477.90 to 5619.80]

22. Primary Outcome: RSV-A Neutralizing Titers for Maternal Participants at Pre-dosing (Day 1)
Description: RSV-A neutralizing titers were determined by neutralization assay and expressed as geometric mean titers (GMTs).
Time Frame: At pre-dosing (Day 1)
Population: as for outcome 20
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | RSV_MAT Group-Mother | Control Group-Mother
Number analyzed (Participants) | 103 | 48
Titers | 681.5 [578.33 to 803.11] | 752.4 [580.25 to 975.50]

23. Primary Outcome: RSV-A Neutralizing Titers for Maternal Participants at Delivery
Description: RSV-A neutralizing titers were determined by neutralization assay and expressed as GMTs.
Time Frame: At delivery
Population: as for outcome 21
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | RSV_MAT Group-Mother | Control Group-Mother
Number analyzed (Participants) | 99 | 44
Titers | 6240.3 [5026.02 to 7747.88] | 612.8 [455.82 to 823.83]

24. Primary Outcome: Geometric Mean Ratio (GMR) Between Cord Blood and Maternal RSV MAT IgG-specific Antibody Concentrations
Description: The placental transfer ratio of IgG-specific antibody concentration was determined from cord blood (or infant blood sample collected within 72 hours after birth [if no cord blood could be obtained]) over that of the blood sample from mother at delivery (if no blood sample was collected during delivery).
Time Frame: At delivery (for maternal participants) or within 72 hours after birth (for infant participants)
Population: Analysis was performed on all pairs of maternal participants (from Per Protocol Set Immunogenicity - Maternal) and their infants (from Per Protocol Set Immunogenicity - Infant) with available results for this outcome measure at the specified time points.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Groups:
- RSV_MAT Group: This group consisted of pairs of maternal participants from RSV_MAT Group - Mother and infant participants from RSV_MAT Group - Infant.
- Control Group: This group consisted of pairs of maternal participants from Control Group - Mother and infant participants from Control Group - Infant.
Arm/Group | RSV_MAT Group | Control Group
Number analyzed (Participants) | 86 | 37
Ratio | 1.33 [1.04 to 1.70] | 2.30 [1.63 to 3.25]

25. Primary Outcome: RSV MAT IgG-specific Antibody Concentrations for Infant Participants at Delivery or Within 72 Hours After Birth
Description: RSV MAT IgG-specific antibody concentrations were determined by ELISA and expressed as GMCs in ELU/mL. The antibody concentrations were measured on the cord blood sample collected at delivery, or on a blood sample collected from the infant within 72 hours after birth (if no cord blood sample could be obtained).
Time Frame: At delivery or within 72 hours after birth
Population: Analysis was performed on the Per Protocol Set Immunogenicity - Infant, which included all infant participants in the Exposed set who had post-delivery/birth immunogenicity data available for the specified analysis at the specified time points, minus those who (a) were born less than 4 weeks post-maternal participant dosing and/ or (b) had protocol deviations that lead to exclusion.
Measure: Geometric Mean (95% Confidence Interval); unit: ELU/mL
Arm/Group | RSV_MAT Group-Infant | Control Group-Infant
Number analyzed (Participants) | 88 | 37
ELU/mL | 77625.1 [63706.97 to 94583.89] | 9228 [6540.47 to 13019.71]

26. Primary Outcome: RSV-A Neutralizing Titers for Infant Participants at Delivery or Within 72 Hours After Birth
Description: RSV-A neutralizing titers were determined by neutralization assay and expressed as GMTs. The titers were measured on the cord blood sample collected at delivery, or on a blood sample collected from the infant within 72 hours after birth (if no cord blood sample could be obtained).
Time Frame: At delivery or within 72 hours after birth
Population: Analysis was performed on the Per Protocol Set Immunogenicity - Infant, which included all infant participants in the Exposed set who had post-delivery/birth immunogenicity data available for the specified analysis at the specified time points, minus those who (a) were born less than 4 weeks post-maternal participant dosing and/ or (b) have protocol deviations that lead to exclusion.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | RSV_MAT Group-Infant | Control Group-Infant
Number analyzed (Participants) | 91 | 37
Titers | 9080.2 [7449.56 to 11067.75] | 694.6 [495.72 to 973.37]

27. Secondary Outcome: Percentage of Maternal Participants Reporting Any SAEs From Day 1 up to 180 Days Post-delivery
Description: as for outcome 4
Time Frame: From Day 1 up to 180 days post-delivery
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RSV_MAT Group-Mother | Control Group-Mother
Number analyzed (Participants) | 113 | 56
Percentage of participants | 29.2 [21.0 to 38.5] | 19.6 [10.2 to 32.4]

28. Secondary Outcome: Number of Maternal Participants Reporting (S)AEs Leading to Study Withdrawal From Day 1 up to 180 Days Post-delivery
Description: as for outcome 5
Time Frame: From Day 1 up to 180 days post-delivery
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | RSV_MAT Group-Mother | Control Group-Mother
Number analyzed (Participants) | 113 | 56
Participants | 0 | 0

29. Secondary Outcome: Percentage of Maternal Participants Reporting MAEs From Day 1 up to 180 Days Post-delivery
Description: as for outcome 13
Time Frame: From Day 1 up to 180 days post-delivery
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RSV_MAT Group-Mother | Control Group-Mother
Number analyzed (Participants) | 113 | 56
Percentage of participants | 61.1 [51.4 to 70.1] | 60.7 [46.8 to 73.5]

30. Secondary Outcome: Percentage of Maternal Participants Reporting Worsening of Pre-existing Medical Conditions and/or Obstetric Complications From Day 1 up to 180 Days Post-delivery
Description: Worsening of pre-existing medical condition and/or obstetric complication was considered by the investigator, using clinical judgement and the following criteria:
  * Change in medication and/or medication dose.
  * Medically attended event in relation to pre-existing condition and/or obstetric complication that are outside the routine management of the condition/complication.
  * SAE and/or hospitalization in relation to pre-existing condition and/or obstetric complication.
Time Frame: From Day 1 up to 180 days post-delivery
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RSV_MAT Group-Mother | Control Group-Mother
Number analyzed (Participants) | 113 | 56
Percentage of participants
  Change In Medication And/Or Medication Dose | 1.8 [0.2 to 6.2] | 1.8 [0.0 to 9.6]
  Medically Attended Event In Relation To Pre-Existing Condition And/Or Obstetric Complication | 1.8 [0.2 to 6.2] | 7.1 [2.0 to 17.3]
  SAE And/Or Hospitalization In Relation To Pre-Existing Condition And/Or Obstetric Complication | 1.8 [0.2 to 6.2] | 3.6 [0.4 to 12.3]

31. Secondary Outcome: Number of Maternal Participants Reporting RSV-associated Medically Attended Respiratory Tract Illnesses (MA-RTIs) From Day 1 up to 180 Days Post-delivery
Description: RSV-associated MA-RTI was defined as a medically attended visit for RTI symptoms and confirmed RSV infection.
Time Frame: From Day 1 up to 180 days post-delivery
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | RSV_MAT Group-Mother | Control Group-Mother
Number analyzed (Participants) | 113 | 56
Participants | 0 | 0

32. Secondary Outcome: Percentage of Infant Participants Reporting Medically Assessed, RSV-associated Lower Respiratory Tract Illness (LRTIs) of Any Severity and RSV-associated Severe LRTIs From Birth up to 365 Days Post-birth
Description: An RSV-associated LRTI is characterized by a history of cough OR difficulty in breathing, AND a blood oxygen saturation by pulse oximetry (SpO2) lower than (<) 95%, OR respiratory rate increase AND a confirmed RSV infection. An RSV-associated severe LRTI meets the case definition of RSV-LRTI AND is additionally characterized by a SpO2 <93%, OR lower chest wall in-drawing, OR inability to feed, OR failure to respond/unconscious.
Time Frame: From birth up to 365 days post-birth
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RSV_MAT Group-Infant | Control Group-Infant
Number analyzed (Participants) | 132 | 66
Percentage of participants
  Any RSV-associated LRTIs | 0.8 [0.0 to 4.1] | 3.0 [0.4 to 10.5]
  RSV-associated Severe LRTIs | 0 [0 to 2.8] | 0 [0 to 5.4]

33. Secondary Outcome: Percentage of Infant Participants Reporting Medically Assessed, RSV-associated Hospitalizations From Birth up to 365 Days Post-birth
Description: RSV-associated hospitalization was defined as a confirmed RSV infection and hospitalized for acute medical condition. Hospitalization was defined as admission for observation or treatment based on the judgment of a health care provider.
Time Frame: From birth up to 365 days post-birth
Population: Analysis was performed on the Exposed Set - Infant, which included infants live-born to exposed maternal participants, whose parents/LARs completed the informed consent process and signed the informed consent.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RSV_MAT Group-Infant | Control Group-Infant
Number analyzed (Participants) | 132 | 66
Percentage of participants | 0.8 [0.0 to 4.1] | 0 [0 to 5.4]

34. Secondary Outcome: RSV MAT IgG-specific Antibody Concentrations for Maternal Participants at Day 31 Post-dosing
Description: RSV MAT IgG-specific antibody concentrations were determined by ELISA and expressed as GMCs in ELU/mL.
Time Frame: At Day 31 post-dosing
Population: Analysis was performed on the Per Protocol Set Immunogenicity - Maternal, which included all maternal participants who received 1 dose of a study intervention and had immunogenicity data available for the specified analysis at the specified time point (i.e. Day 31 post-dosing), minus those participants with protocol deviations that lead to exclusion.
Measure: Geometric Mean (95% Confidence Interval); unit: ELU/mL
Arm/Group | RSV_MAT Group-Mother | Control Group-Mother
Number analyzed (Participants) | 89 | 38
ELU/mL | 113957.1 [102340.44 to 126892.37] | 5510.6 [4370.30 to 6948.51]

35. Secondary Outcome: RSV-A Neutralizing Titers for Maternal Participants at Day 31 Post-dosing
Description: RSV-A neutralizing titers were determined by neutralization assay and expressed as GMTs.
Time Frame: At Day 31 post-dosing
Population: as for outcome 34
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | RSV_MAT Group-Mother | Control Group-Mother
Number analyzed (Participants) | 89 | 38
Titers | 9959.7 [8239.95 to 12038.40] | 575.2 [418.40 to 790.84]

36. Secondary Outcome: RSV-B Neutralizing Titers for Maternal Participants at Pre-dosing (Day 1), Day 31 Post-dosing and Delivery
Description: RSV-B neutralizing titers were determined by neutralization assay and expressed as GMTs.
Time Frame: At pre-dosing (Day 1), Day 31 post-dosing and delivery
Population: Analysis was performed on the Per Protocol Set Immunogenicity - Maternal, which included all maternal participants who received 1 dose of a study intervention and had immunogenicity data available for the specified analysis at the specified time points, minus those participants with protocol deviations that lead to exclusion.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | RSV_MAT Group-Mother | Control Group-Mother
Number analyzed (Participants) | 103 | 47
Titers
  Day 1 | 756.6 [646.03 to 885.98] | 863.4 [664.87 to 1121.12]
  Day 31: number analyzed (Participants) | 89 | 38
  Day 31 | 9928.9 [8331.29 to 11832.87] | 640.7 [475.93 to 862.38]
  Delivery: number analyzed (Participants) | 99 | 43
  Delivery | 6336.9 [5261.95 to 7631.49] | 650.2 [492.25 to 858.82]

37. Secondary Outcome: RSV-B Neutralizing Titers for Infant Participants at Delivery or Within 72 Hours After Birth
Description: RSV-B neutralizing titers were determined by neutralization assay and expressed as GMTs. The titers were measured on the cord blood sample collected at delivery, or on a blood sample collected from the infant within 72 hours after birth (if no cord blood sample could be obtained).
Time Frame: At delivery or within 72 hours after birth
Population: as for outcome 25
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | RSV_MAT Group-Infant | Control Group-Infant
Number analyzed (Participants) | 91 | 37
Titers | 9145.5 [7458.74 to 11213.76] | 779.7 [566.83 to 1072.49]

38. Secondary Outcome: RSV MAT IgG-specific Antibody Concentrations for Infant Participants at Day 43 Post-birth
Description: RSV MAT IgG-specific antibody concentrations were determined by ELISA and expressed as GMCs in ELU/mL.
Time Frame: At Day 43 post-birth
Population: Analysis was performed on a sub-cohort from the Per Protocol Set Immunogenicity - Infant, which included the infant participants for whom blood samples were collected for the specified analysis at Day 43 post-birth.
Measure: Geometric Mean (95% Confidence Interval); unit: ELU/mL
Arm/Group | RSV_MAT Group-Infant | Control Group-Infant
Number analyzed (Participants) | 16 | 5
ELU/mL | 29932.5 [22576.08 to 39686.04] | 1310 [546.48 to 3140.43]

39. Secondary Outcome: RSV MAT IgG-specific Antibody Concentrations for Infant Participants at Day 121 Post-birth
Description: RSV MAT IgG-specific antibody concentrations were determined by ELISA and expressed as GMCs in ELU/mL.
Time Frame: At Day 121 post-birth
Population: Analysis was performed on a sub-cohort from the Per Protocol Set Immunogenicity - Infant, which included the infant participants for whom blood samples were collected for the specified analysis at Day 121 post-birth.
Measure: Geometric Mean (95% Confidence Interval); unit: ELU/mL
Arm/Group | RSV_MAT Group-Infant | Control Group-Infant
Number analyzed (Participants) | 2 | 3
ELU/mL | 4365.1 [12.84 to 1484365.32] | 446.8 [151.14 to 1320.88]

40. Secondary Outcome: RSV MAT IgG-specific Antibody Concentrations for Infant Participants at Day 181 Post-birth
Description: RSV MAT IgG-specific antibody concentrations were determined by ELISA and expressed as GMCs in ELU/mL.
Time Frame: At Day 181 post-birth
Population: Analysis was performed on a sub-cohort from the Per Protocol Set Immunogenicity - Infant, which included the infant participants for whom blood samples were collected for the specified analysis at Day 181 post-birth. There was only one participant in the Control Group - Infant for whom blood sample was collected, hence the 95% confidence interval (CI) associated with geometric mean could not be calculated for single participant.
Measure: Geometric Mean (95% Confidence Interval); unit: ELU/mL
Arm/Group | RSV_MAT Group-Infant | Control Group-Infant
Number analyzed (Participants) | 2 | 1
ELU/mL | 2857.8 [1836.27 to 4447.53] | 241 [NA to NA] — NA indicates that the 95% CI associated with geometric mean could not be calculated for single participant.

41. Secondary Outcome: RSV-A Neutralizing Titers for Infant Participants at Day 43 Post-birth
Description: RSV-A neutralizing titers were determined by neutralization assay and expressed as GMTs.
Time Frame: At Day 43 post-birth
Population: as for outcome 38
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | RSV_MAT Group-Infant | Control Group-Infant
Number analyzed (Participants) | 17 | 5
Titers | 3203.8 [1919.77 to 5346.65] | 240.5 [53.94 to 1072.76]

42. Secondary Outcome: RSV-A Neutralizing Titers for Infant Participants at Day 121 Post-birth
Description: RSV-A neutralizing titers were determined by neutralization assay and expressed as GMTs.
Time Frame: At Day 121 post-birth
Population: as for outcome 39
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | RSV_MAT Group-Infant | Control Group-Infant
Number analyzed (Participants) | 2 | 3
Titers | 607.9 [0.28 to 1322707.87] | 94.1 [68.10 to 130.08]

43. Secondary Outcome: RSV-A Neutralizing Titers for Infant Participants at Day 181 Post-birth
Description: RSV-A neutralizing titers were determined by neutralization assay and expressed as GMTs.
Time Frame: At Day 181 post-birth
Population: as for outcome 40
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | RSV_MAT Group-Infant | Control Group-Infant
Number analyzed (Participants) | 2 | 1
Titers | 755 [0.45 to 1262151.64] | 115 [NA to NA] — NA indicates that the 95% CI associated with geometric mean could not be calculated for single participant.

44. Secondary Outcome: RSV-B Neutralizing Titers for Infant Participants at Day 43 Post-birth
Description: RSV-B neutralizing titers were determined by neutralization assay and expressed as GMTs.
Time Frame: At Day 43 post-birth
Population: as for outcome 38
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | RSV_MAT Group-Infant | Control Group-Infant
Number analyzed (Participants) | 17 | 5
Titers | 3012.8 [1789.81 to 5071.60] | 273.3 [106.14 to 703.45]

45. Secondary Outcome: RSV-B Neutralizing Titers for Infant Participants at Day 121 Post-birth
Description: RSV-B neutralizing titers were determined by neutralization assay and expressed as GMTs.
Time Frame: At Day 121 post-birth
Population: as for outcome 39
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | RSV_MAT Group-Infant | Control Group-Infant
Number analyzed (Participants) | 2 | 3
Titers | 622.7 [2.98 to 129923.70] | 54.9 [27.69 to 108.83]

46. Secondary Outcome: RSV-B Neutralizing Titers for Infant Participants at Day 181 Post-birth
Description: RSV-B neutralizing titers were determined by neutralization assay and expressed as GMTs.
Time Frame: At Day 181 post-birth
Population: as for outcome 40
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | RSV_MAT Group-Infant | Control Group-Infant
Number analyzed (Participants) | 2 | 1
Titers | 327.9 [6.57 to 16367.16] | 63 [NA to NA] — NA indicates that the 95% CI associated with geometric mean could not be calculated for single participant.

ADVERSE EVENTS:
Time Frame: Maternal groups: Solicited AEs - from Day 1 to Day 7 (included) and Unsolicited AEs - from Day 1 to Day 30 (included) after vaccination. SAEs - from Day 1 up to 180 days post-delivery. Infant groups: SAEs and non-serious AEs - from birth up to 365 days post-birth.
Description: "Death neonatal" is considered a serious adverse event for the Control Group-Mother, since the death did not occur from a study pregnancy, but from a subsequent pregnancy. Therefore, due to the fact that the neonate was not considered a study participant, the "death neonatal" event was captured under maternal SAEs.
Arm/Group | RSV_MAT Group-Mother | Control Group-Mother | RSV_MAT Group-Infant | Control Group-Infant
All-Cause Mortality (participants affected / at risk) | 0/113 | 0/56 | 1/132 | 1/66
Serious Adverse Events (participants affected / at risk) | 33/113 | 11/56 | 35/132 | 21/66
Other Adverse Events (participants affected / at risk) | 89/113 | 38/56 | 118/132 | 57/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RSV_MAT Group-Mother (N=113) | Control Group-Mother (N=56) | RSV_MAT Group-Infant (N=132) | Control Group-Infant (N=66)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bradycardia foetal (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Foetal heart rate deceleration abnormality (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary valve stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia foetal (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ankyloglossia congenital (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial septal defect (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Congenital arterial malformation (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Congenital inguinal hernia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cytogenetic abnormality (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fibromatosis colli of infancy (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemangioma congenital (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Newborn persistent pulmonary hypertension (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pectus excavatum (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary valve stenosis congenital (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular septal defect (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intussusception (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Death neonatal (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia neonatal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
ABO incompatibility (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Candida sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysentery (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Endometritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Post procedural cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis neonatal (Infections and infestations) | 0 (0) | 0 (0) | 6 (6) | 3 (3)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Foetal monitoring abnormal (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Medical observation (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia neonatal (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuroblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Poor sucking reflex (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breech delivery (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cephalo-pelvic disproportion (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Failed induction of labour (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Foetal distress syndrome (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Foetal dystocia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Intrapartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 5 (5) | 7 (7)
Low birth weight baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 8 (8) | 4 (4)
Oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Placenta praevia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 7 (7) | 2 (2) | 0 (0) | 0 (0)
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 14 (14) | 5 (5)
Premature labour (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Preterm premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Retained placenta or membranes (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Small for dates baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 3 (3) | 4 (4)
Superimposed pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Threatened labour (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Umbilical cord prolapse (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Vasa praevia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchopulmonary dysplasia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meconium aspiration syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neonatal respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 5 (5) | 2 (2)
Neonatal tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transient tachypnoea of the newborn (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (4) | 2 (2)
Medically induced preterm birth (Surgical and medical procedures) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RSV_MAT Group-Mother (N=113) | Control Group-Mother (N=56) | RSV_MAT Group-Infant (N=132) | Control Group-Infant (N=66)
Nausea (Gastrointestinal disorders) | 28 (28) | 11 (11) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 23 (23) | 10 (10) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 23 (24) | 4 (4) | 6 (6) | 1 (1)
Vomiting (Gastrointestinal disorders) | 9 (9) | 11 (11) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Administration site pain (General disorders) | 50 (50) | 8 (8) | 0 (0) | 0 (0)
Fatigue (General disorders) | 32 (32) | 15 (15) | 0 (0) | 0 (0)
Administration site erythema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Administration site swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site bruising (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 46 (46) | 21 (21) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 4 (5) | 38 (123) | 20 (83)
COVID-19 (Infections and infestations) | 5 (5) | 1 (1) | 4 (4) | 4 (4)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 15 (17) | 7 (11)
Respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 3 (3) | 1 (1)
Bacterial disease carrier (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mastitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 25 (62) | 11 (24)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Premature labour (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Uterine atony (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
False labour (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foetal growth restriction (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foetal hypokinesia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gestational diabetes (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Medically induced preterm birth (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Haematocrit decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Congenital central nervous system anomaly (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 22 (29) | 7 (10)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 6 (8) | 9 (10)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 10 (10) | 3 (5)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 6 (6) | 4 (4)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) | 4 (5)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 5 (8) | 3 (3)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 6 (8) | 2 (2)
Suspected COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 5 (5) | 2 (2)
Otitis media acute (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 3 (4) | 2 (2)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Impetigo (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Candida nappy rash (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Epstein-Barr virus infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tracheobronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Acarodermatitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Body tinea (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bullous impetigo (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coxsackie viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dacryocystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Norovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ophthalmia neonatorum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyoderma (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin candida (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Typhoid fever (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Varicella (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small for dates baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 16 (16) | 14 (14)
Low birth weight baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 17 (17) | 10 (10)
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 10 (10) | 8 (8)
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 7 (7) | 3 (3)
Cephalhaematoma (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Large for dates baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Shoulder dystocia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 10 (11) | 7 (11)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 8 (8) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (4) | 4 (4)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (6)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Acne infantile (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cafe au lait spots (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intertrigo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prurigo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 15 (16) | 9 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 6 (7)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (4) | 2 (2)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Meconium aspiration syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transient tachypnoea of the newborn (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 6 (9) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 4 (4)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Regurgitation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Congenital umbilical hernia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 4 (4) | 4 (4)
Ankyloglossia congenital (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Congenital inguinal hernia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Congenital skin dimples (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cryptorchism (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemangioma congenital (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Naevus flammeus (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Talipes (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (4) | 2 (2)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Weight gain poor (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypoglycaemia neonatal (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lactose intolerance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Underweight (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 2 (4) | 2 (2)
Crying (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Developmental delay (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acquired plagiocephaly (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Joint laxity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint noise (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac murmur (Investigations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Body height below normal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breath sounds abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperbilirubinaemia neonatal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dacryostenosis acquired (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retinopathy of prematurity (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotonia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intraventricular haemorrhage neonatal (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Allergy to arthropod bite (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Milk allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Balanoposthitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Testicular swelling (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrocalcinosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Labial frenectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-03-16): https://cdn.clinicaltrials.gov/large-docs/91/NCT04980391/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-01): https://cdn.clinicaltrials.gov/large-docs/91/NCT04980391/SAP_001.pdf